CLINICAL TRIAL: NCT05924178
Title: A Study on the Effect of Exercise Rehabilitation on Bone Mineral Density, Reconstruction Ligament Tendon Bone Healing and Cartilage After ACL Rupture and Patellar Dislocation
Brief Title: Effects of Preoperative Rehabilitation on Tendon Healing, Bone Mineral Density, and Cartilage After ACLR and Patellar Dislocation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2022837
Record Dates: First submitted 2023-05-28; First posted 2023-06-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-02

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Before ACL reconstruction,40 minutes of rehabilitation training was performed 3 times a week for 6 weeks, and gotted regular treatment. The ACL reconstruction was followed by a 0.5 year rehabilitation.
  Interventions: Behavioral: exercise rehablitation
- control group (Active Comparator): Regular rehabilitation training was not performed before ACL reconstruction, got regular treatment. The ACL reconstruction was followed by a 0.5 year rehabilitation.
  Interventions: Behavioral: routine treatment

INTERVENTIONS:
Behavioral: exercise rehablitation — Preoperative exercise rehabilitation in experimental group was performed.
  Arms: experimental group
Behavioral: routine treatment — The control group receives conventional treatment preoperative.
  Arms: control group

SUMMARY:
To explore the effect of preoperative exercise rehabilitation on bone mineral density, tendon bone healing, change of cartilage, and gait feature in patients with anterior cruciate ligament rupture.

DETAILED DESCRIPTION:
Anterior Cruciate Ligament (ACL) injury is one of the most common sports injuries. It is a serious knee injury. The fracture of ACL can cause functional instability of knee joint, damage of meniscus and articular cartilage, and even induce knee osteoarthritis and other diseases. It has great influence on knee joint and even lower limb function of patients. Arthroscopic ACL reconstruction has become the first choice in clinical treatment of ACL fracture.

ACL fracture can cause local knee joint osteoporosis, and reconstruction surgery can also affect tendon bone healing, bone canal enlargement, rehabilitation period, gait, articular cartilage degradation, etc.

This study intends to conduct preoperative rehabilitation intervention for young people with anterior fork rupture, and explore the effects of exercise rehabilitation on knee bone mineral density, muscle strength, proprioceptive ability and other aspects after ACL rupture, as well as the effects of knee bone mineral density, tendon bone healing, bone tunnel aperture, motor function, gait characteristics and cartilage degradation after reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~40 years old, diagnosed ACL rupture or Patellar Dislocation by MRI;
2. The first unilateral ligamenta reconstruction at our hospital;

Exclusion Criteria:

1. Be older than 40 years, or less than 18 years old
2. Severe injury to other knee ligaments
3. History of knee trauma

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Grade of tendon bone healing | At 6 monthes post operation.
  tendon bone healing by knee MRI
Grade of tendon bone healing | At 1 year post operation.
  tendon bone healing by knee MRI
balanced capacity | At preoperative.
  Y balance test
balanced capacity | At 6 monthes post operation.
  Y balance test
balanced capacity | At 1 year post operation.
  Y balance test
knee T1 rho value | At 6 months post operation.
  knee T1 rho value by functional MRI
knee T1 rho value | At 1 year post operation.
  knee T1 rho value by functional MRI
knee T2 value | At 6 months post operation.
  knee T2 rho value by functional MRI
knee T2 value | At 1 year post operation.
  knee T2 rho value by functional MRI
knee extension angles | At 6 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee extension angles | At 1 year post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
Graft maturity | At 6 monthes post operation.
  tendon bone healing by knee MRI
Graft maturity | At 1 year post operation.
  tendon bone healing by knee MRI
bone mineral density | At preoperative.
  bone mineral density by knee DEX
bone mineral density | At 6 monthes post operation.
  bone mineral density by knee DEX
bone mineral density | At 1 year post operation.
  bone mineral density by knee DEX
isokinetic muscle strength | At preoperative.
  Knee isokinetic strength test
isokinetic muscle strength | At 6 monthes post operation.
  Knee isokinetic strength test
isokinetic muscle strength | At 1 year post operation.
  Knee isokinetic strength test

SECONDARY OUTCOMES:
The HU value of CT | at pre-operation
  CT test

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Can contact the author to communicate and obtain the corresponding data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1/6/2025-1/9/2025
Access Criteria: Relevant data on bone mineral density and physical function can be accessed through the ClinicalTrials.gov website.
URL: http://clinicaltrials.gov/

DOCUMENTS (3):
  • Study Protocol (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT05924178/Prot_001.pdf
  • Statistical Analysis Plan (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT05924178/SAP_002.pdf
  • Informed Consent Form (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT05924178/ICF_003.pdf